CLINICAL TRIAL: NCT07103343
Title: Impact of the MOVI-OLE! [Open Learning Environment] Intervention on Reducing Sedentary Behaviour and Improving Well-being and Cognition in Schools (MOVI-OLE!)
Brief Title: MOVI-OLE! [Open Learning Environments]
Acronym: MOVI-OLE!
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PID2023-148183OB-I00
Record Dates: First submitted 2025-07-19; First posted 2025-08-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Sedentary Behavior; Physical Activity; Cognitive Function; Mental Health; Childhood Obesity; Academic Performance; Executive Function; Health-Related Quality of Life; School Engagement; Cardiometabolic Risk; Classroom Design; Educational Innovation; Physical Fitness; Blood Pressure; Adiposity; Psychological Well-Being
Keywords: Sedentary time; Open Learning Environment; Physical activity; Executive function; Academic achievement; Psychological well-being; Student engagement; Body composition; Adiposity; Cardiorespiratory fitness; Primary school children; Active learning; Educational spaces; Mixed methods
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Psychological Well-Being; Pediatric Obesity; Obesity

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized trial within a parallel design framework.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Classroom (Control Group) (No Intervention): Students in the control group will continue with their usual classroom activities and teaching methodology, without any changes to the furniture or pedagogical approaches during the first year of the study. Teachers in the control group schools will be asked to maintain their standard teaching practices throughout the control period. Traditional classrooms consist of conventional desks and chairs arranged in rows facing the front, with teaching generally teacher-centered. Students usually work individually on assigned tasks.
  For ethical and motivational reasons, this control group will receive the intervention starting in the second academic year.
- MOVI-OLE! -Open Learning Environment- (Intervention Group) (Experimental): Students in the intervention group will experience a classroom environment modified with furniture designed to promote physical activity, alongside the implementation of student-centered teaching methodologies (MOVI-OLE!). Teachers in the intervention group schools will be trained and supported to apply these new methodologies during the school day throughout the study period. The research team will monitor the implementation and provide ongoing assistance to ensure fidelity to the intervention.
  Interventions: Behavioral: MOVI-OLE intervention

INTERVENTIONS:
Behavioral: MOVI-OLE intervention — In the MOVI-OLE! classrooms, traditional desks and chairs will be replaced by three dynamic learning zones:
  A) Dynamic seating: an area with traditional wheeled desks combined with dynamic seats such as fitballs, stools, pedal desks, etc.; B) Standing desks: an area with manually adjustable high desks to allow standing work. Students will also have stools with small backrests and footrests for when they need to sit; C) Vertical boards: vertical boards (vinyl, paper, chalkboard paint, etc.) installed on walls for standing work.
  To facilitate use and adapt to classroom routines, teachers will decide how to distribute students among the different zones, with the requirement that all students spend at least 20 minutes per school day in zone B.
  In addition to the workstations, teachers will receive training and didactic support materials focused on student-centered methodologies and the use of open learning spaces.
  Other Names: MOVI-OLE
  Arms: MOVI-OLE! -Open Learning Environment- (Intervention Group)

SUMMARY:
This study will evaluate the effectiveness of MOVI-OLE! (Open Learning Environment), a school-based intervention designed to reduce sedentary time and enhance multiple aspects of child development, including cognitive function, physical fitness, body composition, psychological well-being, and student engagement. The intervention combines dynamic classroom furniture with student-centered teaching practices. Additionally, a qualitative component will explore how students, teachers, and families perceive the feasibility and acceptability of implementing MOVI-OLE! in real-world school settings.

DETAILED DESCRIPTION:
This study builds on a series of previous school-based interventions (MOVI, MOVI-KIDS, MOVI-da10!, MOVI-HIIT) developed by the research team to promote physical activity and improve health outcomes in children across different educational stages. The new intervention, MOVI-OLE! (Open Learning Environments), aims to address high levels of sedentary behavior during the school day-a growing public health concern associated with poor cardiometabolic health, reduced attention span, and lower psychological well-being in children.

MOVI-OLE! introduces structural and pedagogical changes in the classroom by implementing dynamic learning zones-areas with mobile desks, active seating (e.g., stability balls, stools), standing desks, and wall-mounted writable boards. These physical modifications are supported by teacher training in student-centered pedagogy to promote an active and participatory learning environment.

The intervention will be evaluated through a stepped-wedge cluster randomized controlled trial involving 10 public primary schools in Ciudad Real, Spain. All schools will eventually implement the intervention but in a staggered sequence across two academic years. The primary study population includes students aged 10-12 years (5th and 6th grades of primary education). A pilot phase will precede the main trial to test feasibility and refine procedures.

A mixed-methods approach will be used to assess the impact of the intervention on behavioral, physical, cognitive, emotional, and academic outcomes, as well as to explore perceptions from students, teachers, and families regarding implementation challenges and facilitators.

ELIGIBILITY:
Inclusion Criteria:

* Schools in Ciudad Real (Castilla-La Mancha region) with at least one classroom in both 5rd and 6th grades of Primary Education.
* Schools currently involved in educational innovation projects that aim to transform classrooms and apply student-centered pedagogical approaches.
* Schools whose School Council has approved participation in the MOVI-OLE! intervention and in baseline and final evaluations.
* Students enrolled in 5rd or 6th grade of Primary Education.
* Students without any condition that, according to families, pediatricians, or teachers, prevents participation in the MOVI-OLE! intervention.
* Students with signed informed consent from a parent or legal guardian for participation in the study activities and assessments.
* Students who verbally agree to participate in baseline and final physical assessments.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Sedentary time in classroom | Two academic years
  measured using accelerometers to record sitting/lying, standing, and walking time during classroom activities. Data are expressed as minutes per child during classroom time; higher values of sedentary time indicate greater inactivity.
Sedentary Behavior in Classroom | Two academic years
  measured in a randomly selected subsample using the Portable Ergonomic Observation Method. Observers will record and classify postures (sitting, standing, walking) during classroom time using real-time coding and/or video recordings. Minutes per child per posture category; higher sitting time indicates more sedentary behavior.
Inhibition/Attention | Two academic years
  inhibitory control and attention will be measured using the Flanker Inhibitory Control and Attention Test. Children complete practice trials followed by a block of congruent and incongruent trials. Outcomes include reaction time, accuracy, and raw scores, with higher scores indicating better inhibitory control and attentional performance.
Working memory | Two academic years
  working memory will be assessed using the List Sorting Working Memory Test. Children are required to recall and sequence items presented visually and orally, with task difficulty increasing progressively. Outcomes include raw scores, with higher scores indicating better working memory performance.
Cognitive flexibility | Two academic years
  cognitive flexibility will be assessed using the Dimensional Change Card Sort Test. Children classify stimuli based on color or shape, with blocks assessing both pre-switch and post-switch performance. Outcomes include reaction time, accuracy, and raw scores, with higher scores reflecting greater cognitive flexibility.
Academic performance | Two academic years
  academic grades provided by the school in various subjects, comparing the year prior to the intervention and during the intervention years.
Mental health | Two academic years
  measured with questionnaire such as Revised Children's Anxiety and Depression Scale. This standardized questionnaire assesses a range of anxiety and depression symptoms in children. Responses are rated on a 4-point Likert scale, and scores are converted to age- and sex-normed T-scores. T-scores ≥65 indicate borderline clinical levels, and scores ≥70 indicate clinically significant symptoms.
Health-related quality of life | Two academic years
  measured with questionnaire KIDSCREEN. This standardized instrument evaluates physical, psychological, and social dimensions of well-being in children and adolescents. Items are rated on 5-point Likert scales, and scores are transformed into T-scores. Higher T-scores indicate better HRQoL.
Engagement in the teaching-learning process in students | Two academic years
  student engagement (based on the Achievement Beliefs Scale for Children). This self-report instrument evaluates motivational and cognitive components of academic engagement in children, such as effort, persistence, and beliefs about success. Items are rated on Likert-type scales, with higher scores indicating greater levels of engagement.
Engagement in the teaching-learning process in teachers | Two academic years
  teacher personal efficacy (Utrecht Work Engagement Scale; UWES). This self-report questionnaire measures work engagement through three dimensions: vigor, dedication, and absorption. Items are rated on a 7-point Likert scale. Higher scores indicate greater work engagement and perceived efficacy.
Energy expenditure in classroom in different postures | Two academic years
  estimation of oxigen (O2) consumption during lessons in traditional seated, dynamically seated and standing desks will be assessed in a a randomly selected subsample. It wil be estimated the O2/hour consumption using a K5 COSMED (Oxycon Mobile system; CareFusion) wireless portable metabolic analyzer.

SECONDARY OUTCOMES:
Weight | Two academic years
  weight will be assessed twice using a calibrated digital scale with children barefoot and in lightweight clothing.
Height | Two academic years
  height will be measured twice with a stadiometer, with children standing upright, barefoot, and with the sagittal midline aligned to the wall.
Body mass index (BMI) | Two academic years
  BMI will be calculated as weight divided by height squared (kg/m2).
Body composition | Two academic years
  body compositipon will be assessed twice using the bioimpedance analysis system under standardized conditions (morning, fasting, post-void, after 15 minutes rest, barefoot, with controlled temperature and humidity).
Blood pressure. | Two academic years
  blood pressure will be measured using an automated device (OMRON-M5-I). Systolic and diastolic blood pressure will be assessed twice, with a 5-minute interval between measurements. Children will be seated in a quiet environment, with the right arm semi-flexed at heart level.
Physical activity and sleep | Two academic years
  objectively measured with accelerometers worn for 7 consecutive days, including sleep hours in a subsample.
Cardiorespiratory fitness | Two academic years
  assessed using the 20-meter shuttle run test, which estimates aerobic capacity. Number of completed stages or laps; higher values indicate better fitness.
Muscular Strength | Two academic years
  measured through handgrip strength using a calibrated dynamometer and standing long jump for lower body strength. Handgrip: Kilograms (kg). Horizontal jump: Centimeters (cm).
Speed-Agility | Two academic years
  measured using the 4×10 meter shuttle run test, assessing coordination, speed, and agility. Seconds (s); lower scores indicate better performance.
Self-Reported Neck and Back Pain | Two academic years
  assessed using the Standardized Nordic Musculoskeletal Questionnaire (NMQ), which includes questions about frequency and intensity of neck and back pain over the past 12 months and the past 7 days.Presence of pain (yes/no), and categorical frequency scores (e.g., never, occasionally, often, always); higher values indicate more frequent pain.
Perceptions of the MOVI-OLE! Intervention | Two academic years
  qualitative study will explore the perceptions of teachers, students, and school leadership regarding the facilitators and barriers to implementing the MOVI-OLE! classroom intervention. Data will be collected using qualitative research techniques (e.g., semi-structured interviews, focus groups) and analyzed through thematic analysis. Thematic categories and frequency of themes across stakeholder groups.
Birth and Perinatal Data | Baseline
  collected from parent questionnaires and/or health records. Includes birth weight (kg), gestational age (weeks), breastfeeding status (yes/no), and maternal weight gain during pregnancy (kg). Variable-specific (e.g., kg for weight, weeks for gestational age); categorical for breastfeeding (yes/no).
Parental Weight and BMI | Baseline
  self-reported parental weight and height will be used to calculate Body Mass Index (BMI) for both parents. Weight: kilograms (kg); Height: meters (m); BMI: kg/m2.
Recreational Sedentary Behavior and Screen Time | Baseline
  assessed using parent-reported questionnaires on children's sedentary recreational activities and screen time outside school hours. Minutes per day; higher values indicate more sedentary time.
Eating Habits | Baseline
  dietary intake and food patterns assessed using the Children's Eating Habits Questionnaire (CEHQ). Scale-specific scores; higher values may indicate healthier or unhealthier habits depending on the subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Mairena Sánchez-López, PhD, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- Social and Health Research Center. Universidad de Castilla-La Mancha, Cuenca, Spain

IPD SHARING:
Plan to Share IPD: No